CLINICAL TRIAL: NCT03821324
Title: Clinical Evaluation of the Safety and Performance of Fractional Radiofrequency for the Treatment and Reduction of Acne Scarring
Brief Title: Clinical Evaluation of Fractional Radiofrequency for the Treatment Acne Scarring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Venus Concept (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VI1118
Record Dates: First submitted 2019-01-28; First posted 2019-01-29 (Actual); Results first posted 2023-08-04 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2021-03

CONDITIONS: Acne Scars
Keywords: acne scarring; acne scar; fractional radiofrequency; fractional RF

STUDY DESIGN:
Masking Description: Blinded evaluation of photographs taken at baseline and at 6, 12 weeks post final treatment by independent evaluators.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Intervention (Other): Device: Venus Viva
  Interventions: Device: Venus Viva

INTERVENTIONS:
Device: Venus Viva — The Venus Viva™ fractional RF device has been shown in clinical studies to improve various skin conditions related to aging and alter collagen structures such as wrinkles, rhytids and scars. Beginning with the Baseline visit (Visit 1), subjects will receive a total of 3 treatments approximately 3-5 weeks apart. The left and right side of the face will be treated and assessed as independent sites, and the same applicator tip configuration will be used to treat both sides at all 3 treatment visits.

SUMMARY:
Prospective, single centre, evaluator-blind study of the safety and performance of fractional radiofrequency (RF) for the treatment and reduction of acne scarring. The study will evaluate the progress of 15 subjects requesting treatment of acne scarring. The study will involve three treatments on both sides of the face with 3-5 week intervals between each treatment. Subjects will be followed at 6 and 12 weeks after their last treatment. Analysis will be performed on all subjects who receive at least one treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy, male or female subjects over 21 years of age who are seeking treatment and reduction of their acne scarring.
2. Able to read, understand and voluntarily provide written Informed Consent.
3. Able and willing to comply with the treatment/follow-up schedule and requirements.
4. Women of child-bearing age are required to be using a reliable method of birth control at least 3 months prior to study enrollment and for the duration of the study and have a negative Urine Pregnancy test at baseline.

Exclusion Criteria:

1. Implantable defibrillators, cardiac pacemakers, and other metal implants
2. Subjects with any implantable metal device in the treatment area
3. Pacemaker or internal defibrillator, or any other active electrical implant anywhere in the body (e.g. cochlear implant).
4. Permanent implant in the treated area, such as metal plates and screws, or an injected chemical substance.
5. Current or history of any kind of cancer, or pre-malignant moles.
6. Severe concurrent conditions, such as cardiac disorders.
7. Pregnancy or intending to become pregnant during the study and nursing.
8. Impaired immune system due to immunosuppressive diseases, such as AIDS and HIV, or use of immunosuppressive medications.
9. History of diseases stimulated by heat, such as recurrent herpes simplex in the treatment area; may be enrolled only after a prophylactic regime has been followed for 2 weeks or longer prior to enrollment, or according to Investigator's discretion.
10. Poorly controlled endocrine disorders, such as diabetes.
11. Any active condition in the treatment area, such as sores, psoriasis, eczema, and rash.
12. History of skin disorders, such as keloids, abnormal wound healing, as well as very dry and fragile skin.
13. History of bleeding coagulopathies, or use of anticoagulants (excluding daily aspirin).
14. Facial dermabrasion, facial resurfacing, or deep chemical peeling within the last three months, if face is treated.
15. Use of isotretinoin (Accutane®) or other systemic retinoids within six months or topical retinoids within three months prior to treatment; or as per physician's discretion.
16. Use of non-steroidal anti-inflammatory drugs (NSAIDS, e.g. ibuprofen-containing agents) one week before and after each treatment session.
17. Any surgical procedure in the treatment area within the last six months or before complete healing.
18. Treating over tattoo or permanent makeup.
19. Excessively tanned skin from sun, tanning beds or tanning creams within the last two weeks.
20. As per the practitioner's discretion, refrain from treating any condition which might make it unsafe for the patient.

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-12-11 (Actual); Primary Completion 2019-10-03 (Actual); Study Completion 2019-10-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Gronski, Study Director — Venus Concept
Locations (1):
- Sadick Research Group, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Sides of face
Period: 6 Weeks After Treatment
Arm/Group | Intervention
Started | 14; 28 Sides of face
Completed | 9; 18 Sides of face
Not Completed | 5; 10 Sides of face
Period: 12 Weeks After Treatment
Arm/Group | Intervention
Started | 9; 18 Sides of face
Completed | 9; 18 Sides of face
Not Completed | 0; 0 Sides of face

BASELINE CHARACTERISTICS:
Arm/Group | Intervention
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.5 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 9
  More than one race | 1
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Acne Scar Improvement
Description: Change in acne scarring at 12 weeks post-treatment compared to baseline as assessed by blinded evaluators using photographs a 7-point Global Aesthetic Improvement Scale (GAIS) (ranges from -3 Very Much Worse to +3 Very Much Improved).
Time Frame: 12 weeks post-final treatment (approximately Week 20)
Measure: Mean (Standard Error); unit: units on a scale
Units Other Than Participants: Sides of face
Groups:
- 12-weeks After Last Treatment: Device: Venus Viva
  Venus Viva: The Venus Viva™ fractional RF device has been shown in clinical studies to improve various skin conditions related to aging and alter collagen structures such as wrinkles, rhytids and scars. Beginning with the Baseline visit (Visit 1), subjects will receive a total of 3 treatments approximately 3-5 weeks apart. The left and right side of the face will be treated and assessed as independent sites, and the same applicator tip configuration will be used to treat both sides at all 3 treatment visits.
Arm/Group | 12-weeks After Last Treatment
Number analyzed (Participants) | 9
Number analyzed (Sides of face) | 18
units on a scale | 0.26 (0.12)

2. Secondary Outcome: Subject Satisfaction
Description: Subjects' assessment of satisfaction with the treatment using a 5-point Subject Satisfaction Scale (ranging from 0 Very Unsatisfied to 4 Very Satisfied) at 6 weeks and 12 weeks post-treatment.
Time Frame: 12 weeks post-final treatment (approximately Week 20)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- 12-weeks After Final Treatment: Device: Venus Viva
  Venus Viva: The Venus Viva™ fractional RF device has been shown in clinical studies to improve various skin conditions related to aging and alter collagen structures such as wrinkles, rhytids and scars. Beginning with the Baseline visit (Visit 1), subjects will receive a total of 3 treatments approximately 3-5 weeks apart. The left and right side of the face will be treated and assessed as independent sites, and the same applicator tip configuration will be used to treat both sides at all 3 treatment visits.
Arm/Group | 12-weeks After Final Treatment
Number analyzed (Participants) | 9
units on a scale | 2.89 (1.05)

3. Secondary Outcome: Subject Scale - Visual Analog Scale for Pain
Description: Subjects' assessment of discomfort and pain after treatments as measured by a 10 cm visual analog scale (VAS) with 0 being no pain and 10 being pain as bad as it can be. Each subject was asked to rate their pain after each of the 3 treatments. The result is the mean of each subject's mean VAS score.
Time Frame: Immediately post-treatment at each treatment (average of all 3 treatments)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 14
units on a scale | 3.09 (1.92)

4. Secondary Outcome: Treatment Tolerability
Description: Subjects' assessment of treatment tolerability as measured by a 5-point scale ranging from 0 (Very Intolerable) to 4 (Very Tolerable).
Time Frame: Immediately post-treatment at each treatment (mean of the tolerability scores following each of the 3 treatments)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Intervention: Device: Venus Viva
  Venus Viva: The Venus Viva™ fractional RF device has been shown in clinical studies to improve various skin conditions related to aging and alter collagen structures such as wrinkles, rhytids, and scars. Beginning with the Baseline visit (Visit 1), subjects will receive a total of 3 treatments approximately 3-5 weeks apart. The left and right sides of the face will be treated and assessed as independent sites, and the same applicator tip configuration will be used to treat both sides at all 3 treatment visits.
Arm/Group | Intervention
Number analyzed (Participants) | 14
units on a scale | 3.51 (0.45)

ADVERSE EVENTS:
Time Frame: 5 months
Arm/Group | Intervention
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 3/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=14)
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) — Mild, Probably related
Head Cold (Infections and infestations) | 1 (1) — Mild, Not-related to treatment
Shingles (Infections and infestations) | 1 (1) — Moderate, Not related to treatment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-09): https://cdn.clinicaltrials.gov/large-docs/24/NCT03821324/Prot_SAP_000.pdf